CLINICAL TRIAL: NCT02336971
Title: Individual Prolonged Exposure (PE) Versus Couples' Cognitive-Behavioral Therapy for Combat-Related Posttraumatic Stress Disorder (PTSD)
Brief Title: Individual PE vs Couples' CBT for Combat-Related Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Candice Monson, Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RyersonU
Record Dates: First submitted 2014-12-19; First posted 2015-01-13 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: PTSD; Marital Relationship
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBCT for PTSD (Experimental): CBCT for PTSD is a time-limited, problem-focused treatment that aims to improve PTSD and relationship functioning. The study investigators have developed a 15-session treatment plan each session lasting 75-minutes.
  The treatment is sequenced such that the rationale and psychoeducation provide the basis for the behavioral skills training designed to improve communication and relationship functioning, and to overcome behavioral and experiential avoidance. These skills are used in the final phase of the treatment that is focused on cognitive mechanisms contributing to PTSD and relationship dysfunction.
  Interventions: Behavioral: CBCT for PTSD
- Prolonged Exposure (Experimental): PE for combat-related stress disorders [13-14] serves as the comparison treatment.
  The therapy is usually conducted in 10-12 sessions, each lasting 90-minutes, with the majority of the sessions devoted to imaginal exposure to traumatic memories and homework assignments that include in vivo exposure assignments. In the present study, participants will complete 12 sessions of PE to equate the number of sessions with those of CBCT. Partners of individuals with PTSD are not typically incorporated into the treatment program and so for this study a revised version of PE [1-3] will be administered in which the partner is seen during the second session to discuss PTSD, other reactions to trauma and the treatment procedures.
  Interventions: Behavioral: Prolonged Exposure

INTERVENTIONS:
Behavioral: CBCT for PTSD — CBCT consists of three phases of treatment: Phase 1: treatment orientation and education about PTSD and its related intimate relationship problems Phase 2: behavioral communication skills training Phase 3: cognitive interventions based on Cognitive Processing Therapy (CPT)
  Arms: CBCT for PTSD
Behavioral: Prolonged Exposure — PE consists of: psychoeducation and some limited distress management training, but emphasizes the role of imaginal and in vivo exposure in treating PTSD.
  Arms: Prolonged Exposure

SUMMARY:
This study seeks to enroll 76 couples in which one of the members is a combat-veteran with PTSD. Each couple will be randomized into one of two cognitive-behavioral therapies developed specifically as a treatment for PTSD-either Prolonged Exposure (PE) [1-4] or Cognitive-Behavioral Couples Therapy (CBCT) [5-7]. Whereas, PE was developed as a one-on-one therapy that focuses on treating the individual, CBCT for PTSD incorporates the partners into therapy and seeks to directly address relationship functioning while treating the PTSD symptomatology. Both partners in each couple will complete a battery of several assessments measuring various aspects of psychological distress (e.g., depression, PTSD) and relationship functioning at five time-points throughout the study. But, only the partners assigned to the CBCT group will be involved in the actual therapy sessions. Analysis will be carried out to identify whether any significant differences exist between PE and CBCT in treating PTSD and improving relationship functioning.

DETAILED DESCRIPTION:
The purpose of the proposed study is to examine the effects of Cognitive-Behavioral treatments for PTSD on PTSD symptoms and relationship functioning in active duty military personnel who have recently returned from combat deployment to Operation Enduring Freedom (OEF), Operation Iraqi Freedom (OIF), or Operation New Dawn (OND) and their partners. Research indicates that PTSD is associated with high levels of relationship distress [8-12]. We will compare a treatment specifically designed to incorporate partners, Cognitive-Behavioral Couples Therapy (CBCT), with an established therapy that focuses on treatment of the individual, Prolonged Exposure (PE). CBCT includes techniques designed both to promote support for the traumatized individual and reduce relationship distress; whereas, PE focuses solely on PTSD symptoms and treats only the patient with PTSD. Therefore, we expect to see greater improvement in intimate relationship functioning with CBCT than with PE, while remaining equally effective in reducing PTSD symptomatology. Our specific hypotheses are as follows:

1. Cognitive-Behavioral Couples Therapy (CBCT) and Prolonged Exposure (PE) will be equally effective in reducing PTSD symptoms in a sample of OEF/OIF/OND Veterans, as measured by the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) and the PTSD Checklist - Stressor Specific Version (PCL-S).
2. CBCT for PTSD will be more effective than PE in improving relationship distress in a sample of OEF/OIF/OND Veterans and their partners, as measured by the Couples Satisfaction Index.
3. CBCT for PTSD will have significantly greater impact than PE on measures of relationship functioning (e.g., intimacy, conflict, aggression) in a sample of OEF/OIF/OND Veterans and their partners.

ELIGIBILITY:
Inclusion Criteria:

* • Married or cohabitating couples who have been together the past 3 months in which one partner is an OEF/OIF/OND veteran with PTSD. Diagnosis of PTSD will be determined by the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). The veteran with PTSD must have experienced a Criterion A event that is a specific combat-related event or high magnitude operational experience that occurred during a military deployment in support of OIF/OEF/OND. The diagnosis of PTSD may be indexed to that event or to another Criterion A event.

  * Both individuals must be willing to make a commitment to treatment as prescribed by their randomization in this study.
  * Speak and read English.
  * Be stable for at least 6 weeks on any psychotropic medications either partner may be taking. This criterion is established in order to minimize the likelihood that significant outcome effects may be attributed to changes in psychotropic medications rather than to the treatment protocol.

Exclusion Criteria:

* • Evidence or admission of severe intimate aggression as indicated by a "yes" endorsement to the one-question screen for severe violence items by either member of the couple occurring within the past 6-months.

  * Partner with PTSD symptoms on the Life Events Checklist (LEC), Deployment Risk and Resilience Inventory (DRRI) subscales (if active duty and is a Veteran of deployment), and PTSD CheckList - Stressor Specific (PCL-S) warranting primary treatment for him or herself.
  * Recent initiation of other treatment (i.e., drug/alcohol treatment) or an identified immediate need for other treatment (i.e., severe suicide risk, current alcohol dependence).
  * Current suicidal ideation severe enough to warrant immediate attention (as determined by the Scale for Suicidal Ideation)
  * Alcohol dependence as assessed using the Alcohol Use Disorders Identification Test (AUDIT).
  * Any severe cognitive impairment that precludes retention of session content across sessions or an ongoing psychotic or bipolar disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
PTSD symptoms, as measured by the CAPS and PCL | Post-treatment (approximately 12 weeks)

SECONDARY OUTCOMES:
PTSD symptoms, as measured by the CAPS and PCL | 3, 6 and 12 month follow-ups
Relationship outcomes, as measured by the Couples Satisfaction Index | Post-treatment (approximately 12 weeks), 3, 6 and 12 month follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Candice M Monson, PhD, Principal Investigator — Toronto Metropolitan University
Locations (3):
- United States (3):
  - Fort Hood Military Base, Fort Hood, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Fort Sam Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Background] Foa EB, Rothbaum BO, Riggs DS, Murdock TB. Treatment of posttraumatic stress disorder in rape victims: a comparison between cognitive-behavioral procedures and counseling. J Consult Clin Psychol. 1991 Oct;59(5):715-23. doi: 10.1037//0022-006x.59.5.715. PMID 1955605
- [Background] Foa EB, Dancu CV, Hembree EA, Jaycox LH, Meadows EA, Street GP. A comparison of exposure therapy, stress inoculation training, and their combination for reducing posttraumatic stress disorder in female assault victims. J Consult Clin Psychol. 1999 Apr;67(2):194-200. doi: 10.1037//0022-006x.67.2.194. PMID 10224729
- [Background] Foa EB, Hembree EA, Cahill SP, Rauch SA, Riggs DS, Feeny NC, Yadin E. Randomized trial of prolonged exposure for posttraumatic stress disorder with and without cognitive restructuring: outcome at academic and community clinics. J Consult Clin Psychol. 2005 Oct;73(5):953-64. doi: 10.1037/0022-006X.73.5.953. PMID 16287395
- [Background] Foa EB, Hembree EA, Rothbaum BO. Prolonged exposure therapy for PTSD: Emotional processing of traumatic experiences - therapist guide. 2007. Oxford University Press.
- [Background] Monson CM, Schnurr PP, Stevens SP, Guthrie KA. Cognitive-Behavioral Couple's Treatment for posttraumatic stress disorder: initial findings. J Trauma Stress. 2004 Aug;17(4):341-4. doi: 10.1023/B:JOTS.0000038483.69570.5b. PMID 15462542
- [Background] Monson CM, Rodriguez BF, Warner R. Cognitive-behavioral therapy for PTSD in the real world: do interpersonal relationships make a real difference? J Clin Psychol. 2005 Jun;61(6):751-61. doi: 10.1002/jclp.20096. PMID 15546144
- [Background] Carroll EM, Rueger DB, Foy DW, Donahoe CP Jr. Vietnam combat veterans with posttraumatic stress disorder: analysis of marital and cohabitating adjustment. J Abnorm Psychol. 1985 Aug;94(3):329-37. doi: 10.1037//0021-843x.94.3.329. No abstract available. PMID 4031230
- [Background] Gold JI, Taft CT, Keehn MG, King DW, King LA, Samper RE. PTSD symptom severity and family adjustment among female Vietnam veterans. Military Psychology. 2007;19:71-81.
- [Background] Jordan BK, Marmar CR, Fairbank JA, Schlenger WE, Kulka RA, Hough RL, Weiss DS. Problems in families of male Vietnam veterans with posttraumatic stress disorder. J Consult Clin Psychol. 1992 Dec;60(6):916-26. doi: 10.1037//0022-006x.60.6.916. PMID 1460153
- [Background] MacDonald C, Chamberlain K, Long N, Flett R. Posttraumatic stress disorder and interpersonal functioning in Vietnam War veterans: a mediational model. J Trauma Stress. 1999 Oct;12(4):701-7. doi: 10.1023/A:1024729520686. PMID 10646188
- [Background] Riggs DS, Byrne CA, Weathers FW, Litz BT. The quality of the intimate relationships of male Vietnam veterans: problems associated with posttraumatic stress disorder. J Trauma Stress. 1998 Jan;11(1):87-101. doi: 10.1023/A:1024409200155. PMID 9479678
- [Background] Foa EB, Hembree EA, Dancu CV, Peterson AL, Cigrang JA, Riggs DS. Prolonged exposure treatment for combat-related stress disorders - provider's treatment manual. 2008. Unpublished manual.
- [Background] Nacasch N, Foa EB, Fostick L, Polliack M, Dinstein Y, Tzur D, Levy P, Zohar J. Prolonged exposure therapy for chronic combat-related PTSD: a case report of five veterans. CNS Spectr. 2007 Sep;12(9):690-5. doi: 10.1017/s1092852900021520. PMID 17805215